CLINICAL TRIAL: NCT03130231
Title: The Predictive Value of β2-microspheres for Postoperative Delirium in the Elderly After Orthopedic Surgery
Brief Title: Predictive Value of β2-microspheres for Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian-jun Yang, Director, Department of Anesthesiology, Zhongda Hospital
Other Study IDs: 199101026046
Record Dates: First submitted 2017-04-15; First posted 2017-04-26 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Delirium
Keywords: Delirium β2-microspheres
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: POD group refers to the patients who were diagnosed to be delirious by the Confusion Assessment Method.
- Non-POD group: Non-POD refered to the patients who did not become delirious by the Confusion Assessment Method.

SUMMARY:
This study evaluated the predictive value of β2-microspheres for postoperative delirium (POD) in the elderly after orthopedic surgery. For this purpose, the levels of β2-microspheres in plasma and cerebrospinal fluid were compared between the POD and non-POD groups.

DETAILED DESCRIPTION:
In this study, plasma and cerebrospinal fluid of the patients were collected to detect the levels of β2-microspheres before operation. Also, the patients were interviewed one day before the surgery and on postoperative days 1-3 by the Confusion Assessment Method and then divided them into POD and non-POD groups. The aim of the present study was to assess whether higher levels of β2-microspheres could predict the occurrence of POD.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old, American Standards AssociationⅠ-Ⅲ, undergoing orthopedic operations under spinal anesthesia

Exclusion Criteria:

* decline to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged ≥65 years undergoing orthopedic operations under spinal anesthesia were investigated.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
The incidence of POD | 4 days
  The patients were interviewed one day before the surgery and on postoperative days 1-3 by the Confusion Assessment Method and then divided them into POD and non-POD groups.

SECONDARY OUTCOMES:
The levels of β2-microspheres in plasma and cerebrospinal fluid | 1 day
  Before surgery, plasma and cerebrospinal fluid of the patients were collected to detect the levels of β2-microspheres.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-jun Yang, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No